CLINICAL TRIAL: NCT03568318
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Upadacitinib in Combination With Topical Corticosteroids in Adolescent and Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate Upadacitinib in Combination With Topical Corticosteroids in Adolescent and Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: AD Up
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-047; 2017-005126-37 (EudraCT Number)
Expanded Access: NCT04159597 (Available)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Upadacitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo / Upadacitinib + Topical Corticosteroids (Placebo Comparator): Participants will receive placebo orally once a day (QD) for 16 weeks in the double-blind treatment period. At Week 16 participants will be re-randomized to receive either upadacitinib 15 mg or upadacitinib 30 mg QD up to Week 260. Participants will also receive concomitant topical corticosteroids following a step-down regimen through Week 52.
  Interventions: Drug: Placebo; Drug: Upadacitinib; Drug: Topical corticosteroids (TCS)
- Upadacitinib 15 mg QD + Topical Corticosteroids (Experimental): Participants will receive upadacitinib 15 mg orally once a day for up to 260 weeks. Participants will also receive concomitant topical corticosteroids following a step-down regimen through Week 52.
  Interventions: Drug: Upadacitinib; Drug: Topical corticosteroids (TCS)
- Upadacitinib 30 mg QD + Topical Corticosteroids (Experimental): Participants will receive upadacitinib 30 mg orally once a day for up to 260 weeks. Participants will also receive concomitant topical corticosteroids following a step-down regimen through Week 52.
  Interventions: Drug: Upadacitinib; Drug: Topical corticosteroids (TCS)
- Long-Term Extension (Experimental): Participants who reach Week 260 in Studies M16-045, M18-891, and M16-047 will have the opportunity to roll over into the blinded LTE period of M16-047 to continue receiving the same daily dose of upadacitinib for up to Week 524.
  Interventions: Drug: Upadacitinib; Drug: Topical corticosteroids (TCS)

INTERVENTIONS:
Drug: Placebo — Tablets taken orally once a day
  Arms: Placebo / Upadacitinib + Topical Corticosteroids
Drug: Upadacitinib — Tablets taken orally once a day
  Other Names: ABT-494; RINVOQ™
Drug: Topical corticosteroids (TCS) — Topical corticosteroids will be applied in a stepdown regimen, starting with medium potency once daily to areas with active lesions until lesions are clear or almost clear, or for 3 consecutive weeks, whichever is shorter; then low potency topical corticosteroids once daily. If lesions return or persist, this step-down approach will be repeated until lesion resolution or evidence of local or systemic topical corticosteroids toxicity.
  Recommended TCS include triamcinolone acetonide 0.1% cream or fluocinolone acetonide 0.025% ointment as medium potency topical corticosteroids and hydrocortisone 1% cream as low potency topical corticosteroid.

SUMMARY:
The objective of this study is to assess the efficacy and safety of upadacitinib combined with topical corticosteroids (TCS) for the treatment of adolescent and adult participants with moderate to severe atopic dermatitis (AD) who are candidates for systemic therapy.

DETAILED DESCRIPTION:
This study includes a 35-day screening period, a 16-week double-blind period, a blinded extension period up to Week 260, a blinded Long-term Extension (LTE) Period after Week 260 to Week 524, and a 30-day follow-up visit. Participants who meet eligibility criteria in the Main Study will be randomly assigned in a 1:1:1 ratio to receive upadacitinib 15 mg, upadacitinib 30 mg, or placebo once daily, in combination with topical corticosteroids.

Upon completion of enrollment of 810 participants in the Main Study, a supplemental study will continue to enroll adolescent participants (Adolescent Sub-study) until a total of 180 adolescent participants are enrolled in the overall study (Main Study + Adolescent Sub-study).

Approximately 1000 participants from M16-045 or M18-891 and approximately 500 participants from M16-047 will have the opportunity to enroll into the blinded Long-Term Extension (LTE) period (Week 260 - Week 524) after reaching Week 260 in their respective studies.

Randomization for the Main Study will be stratified by Baseline disease severity (validated Investigator Global Assessment Scale for Atopic Dermatitis [vIGA-AD] score of moderate [3] versus severe [4]), by geographic region (US/Puerto Rico/Canada, Japan, China, and Other), and by age (adolescent [ages 12 to 17] versus adult [ages 18 to 75]). The separate randomization for the Adolescent Sub-study will be stratified by Baseline disease severity (moderate [vIGA-AD 3] versus severe [vIGA-AD 4]) and by geographic region (US/Puerto Rico/Canada and Other).

At Week 16 of both the Main Study and the Adolescent Sub-study, participants in the placebo group will be re-randomized in a 1:1 ratio to receive daily oral doses of upadacitinib 30 mg or upadacitinib 15 mg in the blinded extension period, and participants originally randomized to upadacitinib will continue upadacitinib in the extension period at the same dose. For the Main Study, the re-randomization will be stratified by Eczema Area and Severity Index (EASI) 50 responder status (Yes/No), by geographic region (US/Puerto Rico/Canada, Japan, China, and Other) and by age (adolescent [ages 12 to 17] versus adult [ages 18 to 75]). For the Adolescent Sub-study, the re-randomization will be stratified by EASI 50 responder (Yes/No) and by geographic region (US/Puerto Rico/Canada and Other).

Starting at Week 4, rescue treatment for AD may be provided at the discretion of the investigator if medically necessary The Primary Analysis for the Main Study will be conducted after all ongoing participants have completed Week 16. In addition, a Primary Analysis for the adolescent population (including the adolescent participants from the Main Study and the Adolescent Sub-study) will be conducted after all ongoing adolescent participants have completed Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of ≥ 40 kg at Baseline Visit for participants ≥ 12 and < 18 years of age
* Chronic atopic dermatitis (AD) with onset of symptoms at least 3 years prior to Baseline Visit and subject meets Hanifin and Rajka criteria.
* Active moderate to severe atopic dermatitis defined by Eczema Area and Severity Index (EASI) ≥ 16, validated Investigator's Global Assessment (vIGA) ≥ 3, ≥ 10% of body surface area (BSA) with AD involvement, and weekly average of daily Worst Pruritus numerical rating scale (NRS) ≥ 4.
* Subject has applied a topical emollient (moisturizer) twice daily for at least 7 days before the Baseline Visit.
* Documented history of inadequate response to topical corticosteroids or topical calcineurin inhibitor OR documented systemic treatment for AD within 6 months prior to Baseline Visit

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor
* Unable or unwilling to discontinue current atopic dermatitis (AD) treatments prior to the study
* Requirement of prohibited medications during the study
* Other active skin diseases or skin infections requiring systemic treatment or would interfere with appropriate assessment of atopic dermatitis lesions
* Female subject who is pregnant, breastfeeding, or considering pregnancy during the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1533 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2030-10-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (193):
- United States (59):
  - Total Skin and Beauty Derm Ctr /ID# 200548, Birmingham, Alabama
  - Clinical Research Center AL /ID# 201865, Birmingham, Alabama
  - ACCEL Research Sites /ID# 213364, Birmingham, Alabama
  - Advanced Dermatology and Skin Care Centre /ID# 213550, Mobile, Alabama
  - Alliance Dermatology and MOHs Center, PC /ID#200540, Phoenix, Arizona
  - Arizona Research Center, Inc. /ID# 200546, Phoenix, Arizona
  - Clear Dermatology & Aesthetics Center /ID# 201257, Scottsdale, Arizona
  - University of Arizona /ID# 201059, Tucson, Arizona
  - Bakersfield Derma & Skin Cance /ID# 200892, Bakersfield, California
  - Mosaic Dermatology /ID# 200553, Beverly Hills, California
  - University of California Irvine /ID# 200902, Irvine, California
  - Therapeutics Clinical Research /ID# 200593, San Diego, California
  - Stanford University /ID# 200597, Stanford, California
  - Duplicate_University of Colorado Anchutz Medical Campus /ID# 202822, Aurora, Colorado
  - Colorado Center for Dermatology, PLLC /ID# 203626, Centennial, Colorado
  - Duplicate_Western States Clinical Research, Inc. /ID# 201702, Wheat Ridge, Colorado
  - Dermatology Physicians of Connecticut /ID# 201004, Shelton, Connecticut
  - Clearlyderm Dermatology /ID# 207709, Boca Raton, Florida
  - Skin Care Research, LLC /ID# 200812, Boca Raton, Florida
  - Clinical Research of West Florida, Inc /ID# 203643, Clearwater, Florida
  - Florida Academic Centers Research and Education /ID# 200544, Coral Gables, Florida
  - Tory P Sullivan, MD PA /ID# 201174, North Miami Beach, Florida
  - Park Avenue Dermatology, PA /ID# 201012, Orange Park, Florida
  - Precision Clinical Research /ID# 208734, Sunrise, Florida
  - Advanced Clinical Research at Treasure Valley Dermatology & Skin Cancer Center /ID# 203628, Boise, Idaho
  - Northwestern University Feinberg School of Medicine /ID# 201646, Chicago, Illinois
  - Northshore University Health System Dermatology Clinical Trials Unit /ID# 200556, Skokie, Illinois
  - DuPage Medical Group /ID# 202065, Wheaton, Illinois
  - Deaconess Clinic Downtown /ID# 201001, Evansville, Indiana
  - Indiana University /ID# 200515, Indianapolis, Indiana
  - Epiphany Dermatology of Kansas LLC /ID# 203026, Overland Park, Kansas
  - ORA, Inc. /ID# 202824, Andover, Massachusetts
  - Tufts Medical Center /ID# 200570, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 200545, Boston, Massachusetts
  - Clin Res Inst of Michigan, LLC /ID# 208020, Chesterfield, Michigan
  - Michigan Center for Research Company /ID# 200560, Clarkston, Michigan
  - MediSearch Clinical Trials /ID# 201006, Saint Joseph, Missouri
  - Skin Specialists, PC /ID# 200573, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 200918, Lebanon, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey /ID# 200714, East Windsor, New Jersey
  - Juva Skin and Laser Center /ID# 200997, New York, New York
  - J. Schwartz, MD, PLLC /ID# 202122, Troy, New York
  - Bexley Dermatology Research /ID# 200899, Bexley, Ohio
  - The Ohio State University /ID# 200542, Columbus, Ohio
  - Vital Prospects Clinical Research Institute, PC /ID# 200901, Tulsa, Oklahoma
  - Oregon Dermatology and Research Center /ID# 200601, Portland, Oregon
  - University of Pittsburgh MC /ID# 206057, Pittsburgh, Pennsylvania
  - Rhode Island Hospital /ID# 200566, Providence, Rhode Island
  - AAPRI Clinical Research /ID# 221134, Warwick, Rhode Island
  - Rivergate Dermatology & Skin Care Center /ID# 201698, Goodlettsville, Tennessee
  - Stones River Dermatology /ID# 204962, Murfreesboro, Tennessee
  - Arlington Research Center, Inc /ID# 200559, Arlington, Texas
  - Center for Clinical Studies /ID# 200582, Houston, Texas
  - Progressive Clinical Research /ID# 201582, San Antonio, Texas
  - Center for Clinical Studies - Webster TX /ID# 203186, Webster, Texas
  - Advanced Clinical Research - Woseth Dermatology /ID# 213745, Salt Lake City, Utah
  - Eastern Virginia Med School /ID# 200994, Norfolk, Virginia
  - Dermatology Associates of Seattle /ID# 200717, Seattle, Washington
  - University of Wisconsin - Madison /ID# 204933, Madison, Wisconsin
- Australia (5):
  - St George Dermatology & Skin Cancer Centre /ID# 204788, Kogarah, New South Wales
  - Royal North Shore Hospital /ID# 204639, St Leonards, New South Wales
  - Westmead Hospital /ID# 205682, Westmead, New South Wales
  - Veracity Clinical Research /ID# 204793, Woolloongabba, Queensland
  - Fremantle Dermatology /ID# 205306, Fremantle, Western Australia
- Austria (4):
  - Medizinische Universitaet Innsbruck /ID# 210897, Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 209567, Linz, Upper Austria
  - Kepler Universitaetsklinikum GmbH /ID# 201075, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 201080, Vienna, Vienna
- Belgium (4):
  - UZ Brussel /ID# 203557, Jette, Brussels Capital
  - UCL Saint-Luc /ID# 202028, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Gent /ID# 202030, Ghent, Oost-Vlaanderen
  - IMTR - Grand Hopital de Charleroi /ID# 202029, Loverval
- Canada (17):
  - Kirk Barber Research, CA /ID# 200329, Calgary, Alberta
  - Dermatology Research Institute Inc. /ID# 200341, Calgary, Alberta
  - Alberta DermaSurgery Centre /ID# 205674, Edmonton, Alberta
  - Karma Clinical Trials /ID# 200339, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Resea /ID# 200335, Halifax, Nova Scotia
  - Lynderm Research Inc. /ID# 200338, Markham, Ontario
  - DermEdge Research Inc. /ID# 200337, Mississauga, Ontario
  - The Centre for Clinical Trials /ID# 205404, Oakville, Ontario
  - Angela Montgomery Medicine Professional Corporation /ID# 212653, Ottawa, Ontario
  - SKIN Centre for Dermatology /ID# 200331, Peterborough, Ontario
  - The Center For Dermatology /ID# 205409, Richmond Hill, Ontario
  - Toronto Research Centre /ID# 205411, Toronto, Ontario
  - Research Toronto /ID# 205410, Toronto, Ontario
  - XLR8 Medical Research /ID# 205405, Windsor, Ontario
  - CHU Sainte-Justine /ID# 206013, Montreal, Quebec
  - Centre de recheche dermatologique du Quebec Metropolitain /ID# 205403, Québec, Quebec
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 200330, Saint-Jérôme, Quebec
- China (9):
  - Chinese PLA General Hospital /ID# 206786, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University /ID# 206728, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 206669, Wuhan, Hubei
  - The First Hospital of China Medical University /ID# 209840, Shenyang, Liaoning
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 207132, Hangzhou, Zhejiang
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 207442, Hangzhou, Zhejiang
  - Beijing Friendship Hospital /ID# 207434, Beijing
  - Xiangya Hospital Central South University /ID# 207510, Changsha
  - Huashan Hospital of Fudan University /ID# 207437, Shanghai
- Czechia (4):
  - Fakultni nemocnice Plzen /ID# 202044, Pilsen
  - Sanatorium profesora Arenbergera /ID# 202082, Prague
  - Duplicate_Vseobecna Fakultni Nemocnice /ID# 205248, Prague
  - Vseobecna fakultni nemocnice v Praze /ID# 202045, Prague
- France (5):
  - Chu de Nice-Hopital L'Archet Ii /Id# 205780, Nice, Alpes-Maritimes
  - AP-HM - Hopital de la Timone /ID# 206128, Marseille, Bouches-du-Rhone
  - CHRU Tours - Hopital Gatien de Clocheville /ID# 218209, Tours, Centre-Val de Loire
  - Hopital Saint-Andre /ID# 206129, Bordeaux
  - Polyclinique Courlancy /ID# 201537, Reims
- Germany (10):
  - Universitaetsklinik Heidelberg /ID# 202097, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Frankfurt /ID# 202095, Frankfurt am Main, Hesse
  - Universitaetsklinikum Muenster /ID# 202094, Münster, North Rhine-Westphalia
  - CMS3 Company for Medical Study /ID# 205195, Selters, Rhineland-Palatinate
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 202256, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Bonn /ID# 202092, Bonn
  - TFS Trial Form Support GmbH /ID# 202096, Hamburg
  - Medizinische Hochschule Hannover /ID# 202098, Hanover
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz /ID# 205194, Mainz
  - Klinikum rechts der Isar - Technische Universitaet Muenchen /ID# 202093, Munich
- Greece (6):
  - 401 GSNA - 401 Army General Hospital /ID# 211963, Athens, Attica
  - Children's Hosp P. A. Kyriakou /ID# 217573, Athens, Attica
  - University General Hospital Attikon /ID# 201126, Athens, Attica
  - General Hospital Andreas Syggros /ID# 201123, Athens, Attica
  - Papageorgiou General Hospital Thessaloniki /ID# 202392, Stavroupoli (Thessalonikis), Thessaloniki
  - Thessaloniki Hospital of Skin and Venereal Diseases /ID# 201124, Thessaloniki
- Hong Kong (2):
  - Prince of Wales Hospital /ID# 205152, Hong Kong
  - Queen Mary Hospital /ID# 205146, Hong Kong
- Hungary (5):
  - Oroshazi Korhaz /ID# 203525, Orosháza, Bekes County
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 204144, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont /ID# 201765, Debrecen, Hajdú-Bihar
  - Derma-B Egeszsegugyi es Szolgaltato Kft. /ID# 217866, Debrecen
  - Allergo-Derm Bakos Kft. /ID# 205361, Szolnok
- Ireland (3):
  - St James Hospital /ID# 201118, Dublin, Dublin
  - South Infirmary Victoria University Hospital /ID# 201079, Cork
  - University Hospital Waterford /ID# 201253, Waterford
- Israel (5):
  - Soroka University Medical Center /ID# 206652, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 201611, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 201608, Tel Aviv, Tel Aviv
  - HaEmek Medical Center /ID# 201958, Afula
  - Rabin Medical Center /ID# 201959, Petah Tikva
- Italy (6):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 203014, Rome, Lazio
  - Istituto Clinico Humanitas /ID# 200739, Rozzano, Milano
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 200690, Ancona
  - A.O.U. Policlinico G. Rodolico S.Marco- Presidio G.Rodolico /ID# 200742, Catania
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 200744, Milan
  - Azienda Ospedaliera Universitaria Federico II /ID# 200751, Napoli
- Japan (16):
  - Chukyo Hospital /ID# 202311, Nagoya, Aichi-ken
  - Medical Corporation Matsuo Clinic /ID# 202312, Fukuoka, Fukuoka
  - Hiroshima University Hospital /ID# 201914, Hiroshima, Hiroshima
  - Medical Corporation Kojinkai Sapporo Skin Clinic /ID#258665, Sapporo, Hokkaido
  - Hiramoto skin clinic /ID# 204048, Amagasaki-shi, Hyōgo
  - National Hospital Organization Sagamihara National Hospital /ID# 201658, Sagamihara-shi, Kanagawa
  - Queens Square Medical Center dermatology allergology /ID# 203850, Yokohama, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID#258604, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 201654, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 206322, Sendai, Miyagi
  - Osaka Habikino Medical Center /ID# 204243, Habikino-shi, Osaka
  - Jichi Medical University Hospital /ID# 201913, Shimotsuke-shi, Tochigi
  - Juntendo University Hospital /ID# 202888, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 201711, Hachioji-shi, Tokyo
  - Maruyama Dermatology Clinic /ID# 202350, Koto-ku, Tokyo
  - Yamate Dermatological Clinic /ID# 202130, Shinjuku-ku, Tokyo
- Netherlands (4):
  - Erasmus Medisch Centrum /ID# 202196, Rotterdam, South Holland
  - Academisch Medisch Centrum /ID# 202193, Amsterdam
  - Universitair Medisch Centrum Groningen /ID# 202195, Groningen
  - Universitair Medisch Centrum Utrecht /ID# 202194, Utrecht
- Clinical Trials NZ /ID# 205336, Hamilton, New Zealand
- Norway (4):
  - Haukeland University Hospital /ID# 201152, Bergen, Hordaland
  - Universitetssykehuset N-Norge, Harstad /ID# 201269, Harstad, Troms
  - Universitetssykehuset N-Norge, Tromso /ID# 201270, Tromsø, Troms
  - Rikshospitalet OUS HF /ID# 201271, Oslo
- Puerto Rico (3):
  - Dr. Samuel Sanchez PSC /ID# 202002, Caguas
  - Clinical Research Puerto Rico /ID# 203644, San Juan
  - GCM Medical Group PSC - Hato Rey /ID# 202003, San Juan
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 204372, Banská Bystrica
  - Univerzitna nemocnica Martin /ID# 203851, Martin
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 204240, Nové Zámky
  - Fakultna nemocnica s poliklinikou J.A. Reimana Presov /ID# 204373, Prešov
- Spain (6):
  - Hospital Universitario de Puerto Real /ID# 200875, Puerto Real, Cadiz
  - Hospital General Universitario Alicante /ID# 200873, Alicante
  - Hospital Santa Creu i Sant Pau /ID# 201325, Barcelona
  - Hospital Universitario de la Princesa /ID# 201517, Madrid
  - Hospital Universitario 12 de Octubre /ID# 201135, Madrid
  - Hospital Universitario La Paz /ID# 205438, Madrid
- Sweden (4):
  - Skane University Hospital Lund /ID# 201244, Lund, Skåne County
  - Sahlgrenska University Hospital /ID# 201274, Gothenburg, Västra Götaland County
  - Sodersjukhuset /ID# 201242, Stockholm
  - Karolinska University Hospital /ID# 201243, Stockholm
- United Kingdom (7):
  - Barts Health NHS Trust /ID# 201044, London, London, City of
  - Guy's and St Thomas' NHS Foundation Trust /ID# 201193, London, London, City of
  - Guy's and St Thomas' NHS Foundation Trust /ID# 204642, London, London, City of
  - Oxford University Hospitals NHS Foundation Trust /ID# 202052, Oxford, Oxfordshire
  - NHS Tayside /ID# 202081, Dundee, Scotland
  - NHS Greater Glasgow and Clyde /ID# 201374, Glasgow, Scotland
  - Leeds Teaching Hospitals NHS Trust /ID# 201106, Leeds

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Irvine AD, Prajapati VH, Guttman-Yassky E, Simpson EL, Papp KA, Blauvelt A, Chu CY, Hong HC, Gold LFS, de Bruin-Weller M, Bieber T, Kabashima K, Rosmarin D, Sancho C, Calimlim BM, Grada A, Yang Y, Wu X, Levy G, Raymundo EM, Teixeira HD, Silverberg JI. Efficacy and Safety of Upadacitinib in Patients With Moderate-to-Severe Atopic Dermatitis: Phase 3 Randomized Clinical Trial Results Through 140 Weeks. Am J Clin Dermatol. 2025 Nov;26(6):1003-1016. doi: 10.1007/s40257-025-00975-3. Epub 2025 Sep 3. PMID 40900410
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Paller AS, Mendes-Bastos P, Siegfried E, Eichenfield LF, Soong W, Prajapati VH, Lio P, Simpson EL, Raymundo EM, Suravaram S, Hu X, Yang Y, Huang X, Calimlim BM, Platt AM, Su JC, Zheng M, Yamamoto-Hanada K, Teixeira HD, Irvine AD. Upadacitinib in Adolescents With Moderate to Severe Atopic Dermatitis: Analysis of 3 Phase 3 Randomized Clinical Trials Through 76 Weeks. JAMA Dermatol. 2024 Dec 1;160(12):1304-1313. doi: 10.1001/jamadermatol.2024.3696. PMID 39441580
- [Derived] Silverberg JI, Leshem YA, Calimlim BM, McDonald J, Litcher-Kelly L. Psychometric evaluation of the Worst Pruritus Numerical Rating Scale (NRS), Atopic Dermatitis Symptom Scale (ADerm-SS), and Atopic Dermatitis Impact Scale (ADerm-IS). Curr Med Res Opin. 2023 Oct;39(10):1289-1296. doi: 10.1080/03007995.2023.2251883. Epub 2023 Sep 13. PMID 37691437
- [Derived] Thyssen JP, Thaci D, Bieber T, Gooderham M, de Bruin-Weller M, Soong W, Kabashima K, Barbarot S, Luna PC, Xu J, Hu X, Liu Y, Raymundo EM, Calimlim BM, Nduaka C, Gamelli A, Simpson EL. Upadacitinib for moderate-to-severe atopic dermatitis: Stratified analysis from three randomized phase 3 trials by key baseline characteristics. J Eur Acad Dermatol Venereol. 2023 Sep;37(9):1871-1880. doi: 10.1111/jdv.19232. Epub 2023 Jun 21. PMID 37247226
- [Derived] Paller AS, Ladizinski B, Mendes-Bastos P, Siegfried E, Soong W, Prajapati VH, Lio P, Thyssen JP, Simpson EL, Platt AM, Raymundo EM, Liu J, Calimlim BM, Huang X, Gu Y, Hu X, Yang Y, Su JC, Zheng M, Yamamoto-Hanada K, Teixeira HD, Irvine AD. Efficacy and Safety of Upadacitinib Treatment in Adolescents With Moderate-to-Severe Atopic Dermatitis: Analysis of the Measure Up 1, Measure Up 2, and AD Up Randomized Clinical Trials. JAMA Dermatol. 2023 May 1;159(5):526-535. doi: 10.1001/jamadermatol.2023.0391. PMID 37043227
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Silverberg JI, Simpson EL, Calimlim BM, Litcher-Kelly L, Li X, Sun X, Leshem YA. Determining Severity Strata for Three Atopic Dermatitis Patient-Reported Outcome Questionnaires: Defining Severity Score Ranges for the Worst Pruritus Numerical Rating Scale and the Atopic Dermatitis Symptom and Impact Scales (ADerm-SS and ADerm-IS). Dermatol Ther (Heidelb). 2022 Dec;12(12):2817-2827. doi: 10.1007/s13555-022-00836-5. Epub 2022 Nov 4. PMID 36333616
- [Derived] Mendes-Bastos P, Ladizinski B, Guttman-Yassky E, Jiang P, Liu J, Prajapati VH, Simpson EL, Vigna N, Teixeira HD, Barbarot S. Characterization of acne associated with upadacitinib treatment in patients with moderate-to-severe atopic dermatitis: A post hoc integrated analysis of 3 phase 3 randomized, double-blind, placebo-controlled trials. J Am Acad Dermatol. 2022 Oct;87(4):784-791. doi: 10.1016/j.jaad.2022.06.012. Epub 2022 Jun 15. PMID 35714786
- [Derived] Reich K, Teixeira HD, de Bruin-Weller M, Bieber T, Soong W, Kabashima K, Werfel T, Zeng J, Huang X, Hu X, Hendrickson BA, Ladizinski B, Chu AD, Silverberg JI. Safety and efficacy of upadacitinib in combination with topical corticosteroids in adolescents and adults with moderate-to-severe atopic dermatitis (AD Up): results from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2021 Jun 5;397(10290):2169-2181. doi: 10.1016/S0140-6736(21)00589-4. Epub 2021 May 21. PMID 34023009
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M16-047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 171 clinical sites in 22 countries in the Asia-Pacific region, Europe, Middle East, North America, and Oceania.
  The study included a 16-week double-blind treatment period followed by a blinded extension period (ongoing).
  The first 810 adults and adolescents enrolled constituted the Main Study; additional adolescents were enrolled in the Adolescent Substudy to ensure enrollment of a total of 180 adolescent participants overall.
  Results are reported up to Week 16.
Pre-assignment Details: Participants were randomized equally into 1 of 3 treatment groups, stratified by disease severity (validated Investigator Global Assessment Scale for Atopic Dermatitis [vIGA-AD] moderate [3] vs severe [4]), geographic region (US/Puerto Rico/Canada, Japan, China, and Other), and age (adolescent [ages 12 to 17] vs adult [ages 18 to 75]). Randomization for the adolescent substudy was stratified by disease severity (vIGA-AD 3 vs vIGA-AD 4) and geographic region (US/Puerto Rico/Canada vs Other).
Groups:
- Adults: Placebo + Topical Corticosteroids: Participants ≥ 18 years old received placebo orally once a day (QD) and topical corticosteroids (TCS) following a step-down regimen for 16 weeks in the double-blind treatment period.
- Adults: Upadacitinib 15 mg + Topical Corticosteroids: Participants ≥ 18 years old received upadacitinib 15 mg orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
- Adults: Upadacitinib 30 mg + Topical Corticosteroids: Participants ≥ 18 years old received upadacitinib 30 mg orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
- Adolescents: Placebo + Topical Corticosteroids: Adolescent participants (12 - 17 years old) received placebo orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
- Adolescents: Upadacitinib 15 mg + Topical Corticosteroids: Adolescent participants received upadacitinib 15 mg orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
- Adolescents: Upadacitinib 30 mg + Topical Corticosteroids: Adolescent participants received upadacitinib 30 mg orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
Period: Overall Study
Arm/Group | Adults: Placebo + Topical Corticosteroids | Adults: Upadacitinib 15 mg + Topical Corticosteroids | Adults: Upadacitinib 30 mg + Topical Corticosteroids | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Started (Randomized into study) | 264 | 261 | 260 | 63 | 60 | 60
Received Study Drug | 264 | 261 | 260 | 62 | 60 | 60
Completed (Completed Week 16) | 244 | 249 | 250 | 59 | 58 | 60
Not Completed | 20 | 12 | 10 | 4 | 2 | 0
Not completed — Adverse Event | 3 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 2 | 2 | 1 | 0
Not completed — Other | 3 | 1 | 3 | 0 | 0 | 0
Not completed — Ongoing at Time of Analysis | 5 | 3 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Adults: Placebo + Topical Corticosteroids: Participants ≥ 18 years old received placebo orally once a day (QD) and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Adults: Placebo + Topical Corticosteroids | Adults: Upadacitinib 15 mg + Topical Corticosteroids | Adults: Upadacitinib 30 mg + Topical Corticosteroids | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids | Total
Number analyzed (Participants) | 264 | 261 | 260 | 63 | 60 | 60 | 968
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (14.08) | 35.0 (13.29) | 38.3 (14.82) | 15.1 (1.85) | 15.4 (1.65) | 15.3 (1.86) | 32.8 (15.29)
Age, Customized [Count of Participants; unit: Participants]
  12 - 14 years | 0 | 0 | 0 | 23 | 14 | 21 | 58
  15 - 17 years | 0 | 0 | 0 | 40 | 46 | 39 | 125
  18 - < 40 years | 156 | 176 | 158 | 0 | 0 | 0 | 490
  40 - < 65 years | 94 | 80 | 85 | 0 | 0 | 0 | 259
  ≥ 65 years | 14 | 5 | 17 | 0 | 0 | 0 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 104 | 95 | 36 | 27 | 25 | 388
  Male | 163 | 157 | 165 | 27 | 33 | 35 | 580
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 14 | 7 | 8 | 7 | 72
  Not Hispanic or Latino | 249 | 240 | 246 | 56 | 52 | 53 | 896
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3 | 0 | 0 | 0 | 6
  Asian | 52 | 57 | 58 | 14 | 13 | 6 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 1 | 0 | 0 | 0 | 4
  Black or African American | 15 | 15 | 9 | 5 | 5 | 6 | 55
  White | 196 | 177 | 188 | 44 | 41 | 46 | 692
  More than one race | 0 | 7 | 1 | 0 | 1 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Study Enrollment [Count of Participants; unit: Participants]
  Main Study | 264 | 261 | 260 | 40 | 39 | 37 | 901
  Adolescent Substudy | 0 | 0 | 0 | 23 | 21 | 23 | 67
Geographic Region [Count of Participants; unit: Participants]
  US/Puerto Rico/Canada | 90 | 90 | 89 | 31 | 31 | 31 | 362
  Japan | 18 | 16 | 17 | 0 | 0 | 0 | 51
  China | 16 | 15 | 15 | 2 | 2 | 1 | 51
  Other | 140 | 140 | 139 | 30 | 27 | 28 | 504
Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) [Count of Participants; unit: Participants] — The vIGA-AD was used to assess the severity of atopic dermatitis based on lesion appearance on the following scale:
  * 0-Clear: No inflammatory signs of AD;
  * 1-Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2-Mild: Slight but definite erythema, induration/papulation and/or lichenification. No oozing or crusting;
  * 3-Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4-Severe: Marked erythema, induration/papulation and/or lichenification, oozing or crusting may be present.
  Participants
    3 (Moderate) | 123 | 124 | 123 | 28 | 29 | 29 | 456
    4 (Severe) | 141 | 137 | 137 | 35 | 31 | 31 | 512
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  score on a scale | 30.06 (12.860) | 29.03 (11.925) | 29.68 (11.993) | 30.25 (12.105) | 29.59 (11.683) | 28.68 (10.143) | 29.58 (12.082)
Disease Duration since Diagnosis [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 264 | 261 | 260 | 62 | 60 | 60 | 967
    (all) | 25.986 (15.5650) | 24.511 (14.0363) | 24.617 (16.6107) | 12.315 (4.2769) | 11.370 (5.0674) | 12.244 (3.9262) | 22.584 (14.9374)

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Percentage of Participants Achieving at Least a 75% Reduction in Eczema Area and Severity Index Score (EASI 75) From Baseline at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Time Frame: Baseline and Week 16
Population: The intent-to-treat population for the main study (ITT_M) includes all participants who were randomized in the main study (adults and adolescents). Non-responder imputation incorporating multiple imputation to handle missing data due to coronavirus disease 2019 pandemic (COVID-19) (NRI-C) was used.
  The pre-specified primary analysis included participants enrolled in the main study only; Efficacy analyses of adolescent participants were conducted separately and are reported below.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo + Topical Corticosteroids: Participants received placebo orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
- Upadacitinib 15 mg + Topical Corticosteroids: Participants received upadacitinib 15 mg orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
- Upadacitinib 30 mg + Topical Corticosteroids: Participants received upadacitinib 30 mg orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 304 | 300 | 297
percentage of participants | 26.4 [21.5 to 31.4] | 64.6 [59.1 to 70.0] | 77.1 [72.3 to 81.9]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — The overall type I error rate of the coprimary and all key secondary endpoints for upadacitinib 30 mg was controlled at the 0.05 level using a graphical multiple testing procedure following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 50.6, 95% CI 2-sided [43.8 to 57.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — The overall type I error rate of the coprimary and all key secondary endpoints for upadacitinib 15 mg was controlled at the 0.05 level using a graphical multiple testing procedure following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 38.1, 95% CI 2-sided [30.8 to 45.4] — Response Rate Difference = Upadacitinib - Placebo

2. Primary Outcome: Main Study: Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) of 0 or 1 With a Reduction From Baseline of ≥ 2 Points at Week 16
Description: The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No inflammatory signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 304 | 300 | 297
percentage of participants | 10.9 [7.4 to 14.4] | 39.6 [34.1 to 45.2] | 58.6 [53.0 to 64.2]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 47.6, 95% CI 2-sided [41.1 to 54.0] — Response rate difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 28.5, 95% CI 2-sided [22.1 to 34.9] — Response rate difference = Upadacitinib - Placebo

3. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus Numerical Rating Scale (NRS) at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with Worst Pruritus NRS (weekly average) ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 294 | 288 | 291
percentage of participants | 15.0 [10.9 to 19.0] | 51.7 [46.0 to 57.5] | 63.9 [58.4 to 69.4]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 48.8, 95% CI 2-sided [41.9 to 55.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 36.8, 95% CI 2-sided [29.7 to 43.8] — Response Rate Difference = Upadacitinib - Placebo

4. Secondary Outcome: Main Study: Percentage of Participants Achieving a 90% Reduction From Baseline in EASI Score (EASI 90) at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/ neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 304 | 300 | 297
percentage of participants | 13.2 [9.4 to 17.0] | 42.8 [37.2 to 48.4] | 63.1 [57.6 to 68.6]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 49.9, 95% CI 2-sided [43.3 to 56.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 29.5, 95% CI 2-sided [22.8 to 36.3] — Response Rate Difference = Upadacitinib - Placebo

5. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 4
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 294 | 288 | 291
percentage of participants | 15.0 [10.9 to 19.0] | 52.4 [46.7 to 58.2] | 65.6 [60.2 to 71.1]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 50.6, 95% CI 2-sided [43.8 to 57.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 37.4, 95% CI 2-sided [30.4 to 44.3] — Response Rate Difference = Upadacitinib - Placebo

6. Secondary Outcome: Main Study: Percentage of Participants Achieving an EASI 75 Response at Week 4
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 75 response is defined as at least a 75% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 304 | 300 | 297
percentage of participants | 14.8 [10.8 to 18.8] | 58.7 [53.1 to 64.2] | 72.4 [67.3 to 77.5]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 57.6, 95% CI 2-sided [51.2 to 63.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 43.8, 95% CI 2-sided [37.0 to 50.5] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Main Study: Percentage of Participants Achieving an EASI 75 Response at Week 2
Description: as for outcome 6
Time Frame: Baseline and Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 304 | 300 | 297
percentage of participants | 6.9 [4.1 to 9.8] | 31.0 [25.8 to 36.2] | 44.1 [38.5 to 49.8]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 37.2, 95% CI 2-sided [31.0 to 43.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 24.0, 95% CI 2-sided [18.1 to 29.9] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Main Study: Percentage of Participants Achieving an EASI 90 Response at Week 4
Description: as for outcome 4
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 304 | 300 | 297
percentage of participants | 4.9 [2.5 to 7.4] | 28.3 [23.2 to 33.4] | 43.8 [38.1 to 49.4]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 38.8, 95% CI 2-sided [32.8 to 44.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 23.3, 95% CI 2-sided [17.7 to 28.9] — Response Rate Difference = Upadacitinib - Placebo

9. Secondary Outcome: Main Study: Percentage of Participants Achieving a 100% Reduction From Baseline in EASI Score (EASI 100) at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored from 0 [none], to 3 [severe]) for redness, thickness, scratching, and lichenification.
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  The percentage of participants with an EASI 100 response at Week 16 was pre-specified as a ranked secondary endpoint for participants in the Upadacitinib 30 mg + Topical Corticosteroids group versus Placebo + Topical Corticosteroids group only.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 304 | 300 | 297
percentage of participants | 1.3 [0.0 to 2.6] | 12.0 [8.3 to 15.7] | 22.6 [17.8 to 27.3]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 21.2, 95% CI 2-sided [16.3 to 26.1] — Response Rate Difference = Upadacitinib - Placebo

10. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 1
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 294 | 288 | 291
percentage of participants | 3.1 [1.1 to 5.0] | 12.2 [8.4 to 15.9] | 19.2 [14.7 to 23.8]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 16.2, 95% CI 2-sided [11.3 to 21.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 9.2, 95% CI 2-sided [4.9 to 13.4] — Response Rate Difference = Upadacitinib - Placebo

11. Secondary Outcome: Main Study: Percent Change From Baseline in Worst Pruritus NRS at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores. A negative change from Baseline indicates improvement.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with non-missing Baseline and Week 16 values; missing data were handled using a mixed-effect model with repeated measurements (MMRM) including observed measurements at all visits, except that measurements after any rescue medication were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 184 | 260 | 247
percent change | -25.07 [-31.64 to -18.49] | -58.14 [-64.24 to -52.05] | -66.85 [-72.99 to -60.72]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority — The overall type I error rate of the coprimary and all key secondary endpoints for upadacitinib 30 mg was controlled at the 0.05 level using a graphical multiple testing procedure following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, Baseline vIGA-AD category and age in the model; Least Squares (LS) Mean Difference = -41.79, 95% CI 2-sided [-50.46 to -33.11], Standard Error of Mean 4.417 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — The overall type I error rate of the coprimary and all key secondary endpoints for upadacitinib 15 mg was controlled at the 0.05 level using a graphical multiple testing procedure following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 11, analysis 1]; LS Mean Difference = -33.08, 95% CI 2-sided [-41.72 to -24.44], Standard Error of Mean 4.403 — Difference = Upadacitinib - Placebo

12. Secondary Outcome: Main Study: Percent Change From Baseline in EASI Score at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1)] moderate [2], or severe [3]) for Redness (erythema, inflammation), Thickness (induration, papulation, swelling - acute eczema), Scratching (excoriation), and Lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo + Topical Corticosteroids | Upadacitinib 15 mg + Topical Corticosteroids | Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 206 | 275 | 276
percent change | -45.86 [-50.09 to -41.63] | -77.99 [-81.87 to -74.10] | -87.31 [-91.20 to -83.41]
Statistical Analysis 1: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 30 mg + Topical Corticosteroids; The overall type I error rate of the coprimary and all key secondary endpoints for upadacitinib 30 mg was controlled at the 0.05 level using a graphical multiple testing procedure following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for EU/EMA regulatory purposes only; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 11, analysis 1]; LS Mean Difference = -41.45, 95% CI 2-sided [-46.68 to -36.22], Standard Error of Mean 2.662 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + Topical Corticosteroids vs Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority — The overall type I error rate of the coprimary and all key secondary endpoints for upadacitinib 15 mg was controlled at the 0.05 level using a graphical multiple testing procedure following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for EU/EMA regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 11, analysis 1]; LS Mean Difference = -32.13, 95% CI 2-sided [-37.35 to -26.91], Standard Error of Mean 2.659 — Difference = Upadacitinib - Placebo

13. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 75 Response at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: The ITT population for adolescents (ITT_A) consists of all adolescent participants who were randomized in the main study or the adolescent sub-study. Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adolescents: Placebo + Topical Corticosteroids: Adolescent participants received placebo orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 63 | 60 | 60
percentage of participants | 30.3 [18.9 to 41.6] | 63.3 [51.1 to 75.5] | 84.3 [74.9 to 93.6]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 53.1, 95% CI 2-sided [38.8 to 67.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 32.7, 95% CI 2-sided [16.3 to 49.0] — Response Rate Difference = Upadacitinib - Placebo

14. Secondary Outcome: Adolescents: Percentage of Participants Achieving a vIGA-AD of 0 or 1 With a Reduction From Baseline of ≥ 2 Points at Week 16
Description: The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, possible oozing or crusting;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; possible oozing or crusting.
Time Frame: Baseline and Week 16
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 63 | 60 | 60
percentage of participants | 11.2 [3.4 to 19.1] | 38.3 [26.0 to 50.6] | 67.4 [55.5 to 79.4]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 55.4, 95% CI 2-sided [41.4 to 69.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 26.3, 95% CI 2-sided [12.1 to 40.4] — Response Rate Difference = Upadacitinib - Placebo

15. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Worst pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with Worst Pruritus NRS (weekly average) ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 61 | 57 | 56
percentage of participants | 21.3 [11.0 to 31.6] | 45.6 [32.7 to 58.5] | 51.8 [38.7 to 64.9]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 30.5, 95% CI 2-sided [14.1 to 46.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 24.5, 95% CI 2-sided [8.2 to 40.8] — Response Rate Difference = Upadacitinib - Placebo

16. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 90 Response at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 90 response is defined as at least a 90% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 63 | 60 | 60
percentage of participants | 20.7 [10.7 to 30.7] | 48.3 [35.7 to 61.0] | 73.6 [62.3 to 84.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 52.0, 95% CI 2-sided [37.3 to 66.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 27.1, 95% CI 2-sided [11.1 to 43.1] — Response Rate Difference = Upadacitinib - Placebo

17. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 4
Description: as for outcome 15
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 4
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 61 | 57 | 56
percentage of participants | 23.0 [12.4 to 33.5] | 45.6 [32.7 to 58.5] | 46.4 [33.4 to 59.5]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 23.5, 95% CI 2-sided [6.9 to 40.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 22.7, 95% CI 2-sided [6.2 to 39.2] — Response Rate Difference = Upadacitinib - Placebo

18. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 75 Response at Week 4
Description: as for outcome 6
Time Frame: Baseline and Week 4
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 63 | 60 | 60
percentage of participants | 28.6 [17.4 to 39.7] | 54.9 [42.3 to 67.5] | 78.3 [67.9 to 88.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 49.3, 95% CI 2-sided [34.1 to 64.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 26.2, 95% CI 2-sided [9.4 to 43.1] — Response Rate Difference = Upadacitinib - Placebo

19. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 75 Response at Week 2
Description: as for outcome 6
Time Frame: Baseline and Week 2
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 63 | 60 | 60
percentage of participants | 9.5 [2.3 to 16.8] | 33.7 [21.7 to 45.8] | 51.7 [39.0 to 64.3]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 41.5, 95% CI 2-sided [27.8 to 55.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 24.4, 95% CI 2-sided [10.3 to 38.4] — Response Rate Difference = Upadacitinib - Placebo

20. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 90 Response at Week 4
Description: as for outcome 16
Time Frame: Baseline and Week 4
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 63 | 60 | 60
percentage of participants | 9.5 [2.3 to 16.8] | 34.2 [22.1 to 46.3] | 45.0 [32.4 to 57.6]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 34.9, 95% CI 2-sided [20.6 to 49.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 24.5, 95% CI 2-sided [10.4 to 38.7] — Response Rate Difference = Upadacitinib - Placebo

21. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 100 Response at Week 16
Description: EASI is used to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. and the severity score is calculated as the sum of the intensity scores (scored from 0 [none], to 3 [severe]) for redness, thickness, scratching, and lichenification.
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 100 response is defined as a 100% reduction (improvement) from Baseline in EASI score.
  The percentage of participants with an EASI 100 response at Week 16 was pre-specified as a secondary endpoint for participants in the Upadacitinib 30 mg + TCS group versus Placebo + TCS group only.
Time Frame: Baseline and Week 16
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 63 | 60 | 60
percentage of participants | 4.8 [0.0 to 10.0] | 13.3 [4.7 to 21.9] | 25.0 [14.0 to 36.0]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 19.8, 95% CI 2-sided [7.8 to 31.8] — Response Rate Difference = Upadacitinib - Placebo

22. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 1
Description: as for outcome 15
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 1
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 61 | 57 | 56
percentage of participants | 9.8 [2.4 to 17.3] | 8.8 [1.4 to 16.1] | 16.1 [6.5 to 25.7]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p = 0.306, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 6.2, 95% CI 2-sided [-5.7 to 18.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.855, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = -1.0, 95% CI 2-sided [-11.2 to 9.3] — Response Rate Difference = Upadacitinib - Placebo

23. Secondary Outcome: Adolescents: Percent Change From Baseline in Worst Pruritus NRS at Week 16
Description: as for outcome 11
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with non-missing Baseline and Week 16 values; missing data were handled using a mixed-effect model with repeated measurements including observed measurements at all visits, except that measurements after any rescue medication were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 41 | 50 | 49
percent change | -32.96 [-49.87 to -16.05] | -59.34 [-75.78 to -42.90] | -49.02 [-65.35 to -32.69]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p = 0.180, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, and Baseline vIGA-AD category in the model; LS Mean Difference = -16.05, 95% CI 2-sided [-39.59 to 7.48], Standard Error of Mean 11.956 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p = 0.029, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 23, analysis 1]; LS Mean Difference = -26.38, 95% CI 2-sided [-49.97 to -2.79], Standard Error of Mean 11.986 — Difference = Upadacitinib - Placebo

24. Secondary Outcome: Adolescents: Percent Change From Baseline in EASI Score at Week 16
Description: as for outcome 12
Time Frame: Baseline and Week 16
Population: as for outcome 23
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
Number analyzed (Participants) | 48 | 55 | 58
percent change | -53.53 [-61.23 to -45.82] | -77.90 [-85.36 to -70.44] | -89.22 [-96.49 to -81.95]
Statistical Analysis 1: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 30 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 23, analysis 1]; LS Mean Difference = -35.69, 95% CI 2-sided [-46.28 to -25.11], Standard Error of Mean 5.354 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo + Topical Corticosteroids vs Adolescents: Upadacitinib 15 mg + Topical Corticosteroids; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 23, analysis 1]; LS Mean Difference = -24.37, 95% CI 2-sided [-35.10 to -13.65], Standard Error of Mean 5.423 — Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 16, or 30 days after last dose for participants who did not enter the blinded extension period.
Groups:
- Adults: Placebo + Topical Corticosteroids: Participants ≥ 18 years old received placebo orally once a day and topical corticosteroids following a step-down regimen for 16 weeks in the double-blind treatment period.
Arm/Group | Adults: Placebo + Topical Corticosteroids | Adults: Upadacitinib 15 mg + Topical Corticosteroids | Adults: Upadacitinib 30 mg + Topical Corticosteroids | Adolescents: Placebo + Topical Corticosteroids | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids
All-Cause Mortality (participants affected / at risk) | 0/264 | 0/261 | 0/260 | 0/62 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 9/264 | 7/261 | 4/260 | 0/62 | 1/60 | 0/60
Other Adverse Events (participants affected / at risk) | 99/264 | 111/261 | 123/260 | 21/62 | 24/60 | 32/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults: Placebo + Topical Corticosteroids (N=264) | Adults: Upadacitinib 15 mg + Topical Corticosteroids (N=261) | Adults: Upadacitinib 30 mg + Topical Corticosteroids (N=260) | Adolescents: Placebo + Topical Corticosteroids (N=62) | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids (N=60) | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids (N=60)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHEGMATOGENOUS RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULAR STENT THROMBOSIS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONSILLAR ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STATUS ASTHMATICUS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHRODERMIC ATOPIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults: Placebo + Topical Corticosteroids (N=264) | Adults: Upadacitinib 15 mg + Topical Corticosteroids (N=261) | Adults: Upadacitinib 30 mg + Topical Corticosteroids (N=260) | Adolescents: Placebo + Topical Corticosteroids (N=62) | Adolescents: Upadacitinib 15 mg + Topical Corticosteroids (N=60) | Adolescents: Upadacitinib 30 mg + Topical Corticosteroids (N=60)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 6 (7) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 10 (10) | 9 (10) | 4 (4) | 1 (2) | 3 (3)
VOMITING (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
PYREXIA (General disorders) | 3 (3) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 4 (5)
NASOPHARYNGITIS (Infections and infestations) | 31 (38) | 31 (38) | 37 (42) | 3 (3) | 6 (8) | 3 (3)
ORAL HERPES (Infections and infestations) | 5 (7) | 9 (13) | 22 (26) | 1 (1) | 2 (2) | 1 (1)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 1 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 21 (24) | 20 (21) | 19 (21) | 1 (1) | 1 (1) | 4 (7)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 5 (6) | 3 (3) | 1 (1) | 0 (0) | 3 (4)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 7 (7) | 12 (12) | 16 (16) | 1 (1) | 1 (1) | 3 (3)
HEADACHE (Nervous system disorders) | 12 (13) | 11 (13) | 11 (15) | 4 (5) | 5 (5) | 4 (4)
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 10 (11) | 10 (10) | 0 (0) | 3 (3) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 6 (6) | 25 (27) | 36 (39) | 1 (1) | 8 (9) | 9 (9)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 18 (19) | 8 (8) | 2 (2) | 4 (5) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT03568318/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT03568318/SAP_001.pdf